CLINICAL TRIAL: NCT06177873
Title: Effect of Foot Bath on Pain, Anxiety, Sleep and Comfort Level: Randomized Control
Brief Title: Effect of Foot Bath on Pain, Anxiety, Sleep and Comfort Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilek GÜRÇAYIR (Other)
Responsible Party: Sponsor-Investigator, Dilek GÜRÇAYIR, Assistant professor, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 501100004951
Record Dates: First submitted 2023-11-28; First posted 2023-12-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: foot bath; pain; anxiety; comfort; sleep
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Hot water foot bath will applied to intervention group.
  Interventions: Other: foot bath
- control group (No Intervention): Patients in the control group will not have a hot water foot bath and the scales will be applied at the same hours as the patients in the experimental group.

INTERVENTIONS:
Other: foot bath — On the morning of surgery, the purpose of the study will be explained to the patients and their written consent will be obtained. Then, Introductory Information Form, STAI and VASS were applied. The pain level of the patients will be evaluated with VAS-Pain 4 hours after the surgery. SAI and VAS-Comfort will be applied to patients with pain level 4 and above. Then, patients in the experimental group will receive a hot water foot bath for 20 minutes. Before the hot water foot bath, patients will be lifted from their beds and placed on the chair in the room. Hot water will be poured into the foot bath tub and the patient will be asked to put his feet in the water. The water level will be adjusted to include the patients ankles. The temperature of the water will be constantly checked with a water thermometer and kept at 41-42 °C. A hot water foot bath will be applied for 20 minutes and then the patients feet will be dried with a towel.
  Arms: intervention group

SUMMARY:
This study was planned and will conducted to determine the effect of hot foot bath on pain, anxiety, sleep and comfort levels in patients undergoing laparoscopic cholecystectomy.

Research hypotheses H1: A hot foot bath reduces postoperative pain in patients undergoing laparoscopic cholecystectomy.

H2: A hot foot bath reduces postoperative anxiety in patients undergoing laparoscopic cholecystectomy.

H3: A hot foot bath improves postoperative sleep in patients undergoing laparoscopic cholecystectomy.

H4: A hot foot bath improves postoperative comfort in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Nurses play an important role in patients; pain management during the peroperative period. In this process, non-steroidal anti-inflammatory drugs, opioids, patient-controlled analgesia and local anesthetics can be used pharmacologically in pain management. However, it has been reported in the literature that using pharmacological and non-pharmacological applications together in pain management has better positive effects on the patient. Hot application, cold application, transcutaneous electrical nerve stimulation, massage, reiki, music therapy, aromatherapy are some of the non-pharmacological applications used to relieve pain in the postoperative period.

Hot application is one of the effective, cheap and easy-to-use non-pharmacological methods in relieving pain. Hot applications can be made as dry hot, local wet and general wet applications. Foot bath with hot water is one of the non-pharmacological methods that nurses can apply to relieve post-operative patients; pain, reduce anxiety and stress levels, relax muscles and improve sleep quality. There are studies in the literature showing that heat application reduces pain levels and improves sleep quality in different patient groups. In the study of Aghamohammadi et al., it was found that a 20-minute hot foot bath applied to women in menopause improved sleep quality. In the study of Han et al., it was found that hot foot bath with aromatherapy applied to patients with edema in the lower extremities significantly reduced pain and edema. In the study of Soonyoung and Myoungjin, it was determined that hot water foot bath applied to patients who underwent hand replantation reduced the pain of the patients. In another study, hand and foot baths after cesarean section were effective in reducing the pain of patients. When the literature was examined, no study was found examining the effect of hot foot bath on anxiety, pain, sleep and comfort levels after laparoscopic cholecystectomy. In this context, this study was planned and conducted to determine the effect of hot foot bath on pain, anxiety, sleep and comfort levels in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients did not have any psychological disorders, cancer, hypertension or heart disease and did not use any medication related to these diseases
* Patients used the same type of analgesic for pain control in the postoperative period,
* Patients had a VAS pain level of 4 or above, had no foot pain
* Patients who did not have wounds, infections or infectious diseases
* Patients who did not develop any complications before, during and after surgery were

Exclusion Criteria:

* Patients who developed any complications before, during or after surgery
* Patients who had drains were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog pain scale | 4 hours after the surgery, after the application at the 5th, 30th, 60th and 120th minutes.
  Zero is equivalent to no pain and 10 indicates the worst possible pain.
Visual Analog Comfort scale | 4 hours after the surgery, after the application at the 5th, 30th, 60th and 120th minutes.
  Zero is equivalent to no comfort and 10 indicates the worst possible comfort.
Visual Analog Sleep Scale | On the surgery morning, first day after surgery.
  Zero is equivalent to the best sleep and 1000 indicates the worst possible sleep.
The State-Trait Anxiety Inventory Form (STAI) | 4 hours after the surgery, after the application at the 5th, 30th, 60th and 120th minutes.
  20 is equivalent to no anxiety and 80 indicates the worst possible anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No